CLINICAL TRIAL: NCT05868499
Title: Long Term Follow-up Study in Patients With Telomere Biology Disorders With Bone Marrow Failure Who Completed Study EXG-US-01
Brief Title: Rollover Study From EXG-US-01
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Elixirgen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EXG-US-02
Record Dates: First submitted 2023-05-08; First posted 2023-05-22 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Telomere Biology Disorders With Bone Marrow Failure

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EXG34217 (Experimental): single autologous CD34+ cells contacted ex vivo with EXG-001
  Interventions: Biological: EXG34217

INTERVENTIONS:
Biological: EXG34217 — Single infusion

SUMMARY:
This is a long-term rollover follow-up study for Phase I/II study (Protocol EXG-US-01).

DETAILED DESCRIPTION:
Patients who received EXG34217 treatment and had at least one follow-up visit (Month 1, 3, 6, or 12) in Study EXG-US-01 will be eligible for this rollover study. Patient will sign a consent form prior to any study related procedure. This study is to add additional follow-up assessments up to 6 years after EXG34217 treatment. This study does not have additional intervention. Additional visits will be every 6 months in the first 3 years and once a year for two years.

ELIGIBILITY:
Inclusion Criteria:

1. Signed an Institutional Review Board (IRB) approved informed consent document indicating that they understand the purpose of, and procedures required by the study and are willing to participate in the study and comply with all study procedures and restrictions. Informed consent must be obtained from the subject prior to initiating procedures.
2. Have completed the 12-month visit of Study EXG-US-01.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events -Safety by Incidence of Treatment-Emergent | Change from Baseline Systolic Blood Pressure at Month 18, 24,30,36,42,48,60 and 72
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03. Incidence and nature of adverse events, vital signs, weight.
umber of participants with a change in in physical examination | Change from Baseline Systolic Blood Pressure at Month 18, 24,30,36,42,48,60 and 72
  Physical examination changes General appearance ,Head, eyes, ears, nose, and throat, Respiratory, Cardiovascular, Musculoskeletal, Abdomen, Neurologic, Extremities, Dermatologic, Lymphatic)
Number of participants with a change in Electrocardiography (ECG) | Change from Baseline Systolic Blood Pressure at Month 18, 24,30,36,42,48,60 and 72
  ECG (standard digital 12-lead in singlicate)
Number of participants with a change in clinical laboratory evaluations | Change from Baseline Systolic Blood Pressure at Month 18, 24,30,36,42,48,60 and 72
  Changes in clinical laboratory evaluations (Hematology, Blood chemistry, Coagulation, and Urinalysis)
Number of participants with a change of Immunogenicity | Change from Baseline Systolic Blood Pressure at Month 18, 24,30,36,42,48,60 and 72
  Change in Antibody against virus vector and transgene

SECONDARY OUTCOMES:
Number of participants with a change in telomere length | Change from Baseline Systolic Blood Pressure at Month 18, 24,30,36,42,48,60 and 72
  Change in telomere length in any peripheral blood cells
Number of participants with improvement of blood counts. | Change from Baseline Systolic Blood Pressure at Month 18, 24,30,36,42,48,60 and 72
  Blood counts: neutrophils,platelets, or hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Kasiani Myers, MD, Principal Investigator — Cincinnati Children Hospital Medical Center
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States